CLINICAL TRIAL: NCT02679794
Title: Impact of Egg Consumption on Carotenoid and Vitamin D Bioavailability in Pre- and Post-menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph.D., Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1507016290
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Egg consumption (Experimental): Consuming sautéed vegetables and 3g canola oil with 100g (2 large eggs) of whole eggs
  Interventions: Behavioral: Egg consumption
- Control (Placebo Comparator): Consuming sautéed vegetables and 3g canola oil without eggs
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Egg consumption — Subjects will consume a carefully portioned sautéed vegetables and 3g canola oil with 100g (2 large eggs) of whole eggs
  Arms: Egg consumption
Behavioral: Control — Subjects will consume a carefully portioned sautéed vegetables and 3g canola oil.
  Arms: Control

SUMMARY:
The 2010 Dietary Guidelines for Americans emphasizes consumption of 4.5 cups of fruits and vegetables daily but the average intake of US adults is only 2.6 cups. This low consumption of fruits and vegetables results in a limited availability of certain nutrients found in these foods such as carotenoids. Dietary carotenoids have health-promoting properties and are known to fight against disease. Although, maintaining adequate vitamin D status is critical for overall skeletal health and the prevention of osteoporosis, vitamin D insufficiency is also widespread in the United States. Eggs, egg yolk in particular, are known to be a good source of lipid and may improve the absorption of carotenoids and vitamin D found in co-consumed vegetables in young and older women. Therefore, the investigators are interested to see if consuming eggs with cooked vegetables will increase carotenoids and vitamin D absorption.

DETAILED DESCRIPTION:
The 2010 Dietary Guidelines for Americans emphasizes consumption of 4.5 cups of fruits and vegetables daily. However, US adults only consume on average 2.6 cups of fruits and vegetables daily. This low consumption may further result in the limited availability of fat soluble, health-promoting, phytochemicals such as carotenoids (CAT) from these foods. Dietary CAT have beneficial biological properties including antioxidant and anti-inflammatory effects and scientific research supports the protective effects of CAT against many degenerative diseases, including cardiovascular diseases, age-related macular degeneration, and some types of cancer. Therefore, either low intake or inefficient bioavailability of CAT from fruits and vegetables may reduce their potential effectiveness to retard or prevent disease. Recently completed randomized and crossover study found that co-consuming 150g (3 eggs) of scrambled whole eggs (SWE) which contains18g of lipid, increases overall CAT absorption from a mixed-vegetable salad >7-fold compared to a the same salad without eggs (3g of co-consumed lipid) in young healthy men. However, the occurrence of this benefit in women and older adults is unknown. Aging may affect CAT bioavailability due to age-induced physiological changes including reduced gastrointestinal tract function and modifications of chylomicron metabolism. Eggs are known to be a highly bioavailable source of CAT, presumably due to the presence of lipid and phospholipid in egg yolk. The highly bioavailable nature of CAT from eggs suggest that egg-derived factors may be leveraged to improve bioavailability of other CAT found in co-consumed vegetables. While promising, very limited data exist on the impact of a co-consumed food source of lipid to enhance CAT absorption in women or in older adults.

Vitamin D (VIT D) insufficiency is widespread with nearly 2/3 of Americans not meeting the current Institute of Medicine (IOM) recommendation for serum 25-hydroxyvitamin D (25(OH)D) concentration. VIT D has an essential function to regulate calcium homeostasis, including stimulating calcium's active intestinal absorption and renal excretion. Thus, maintaining adequate VIT D status is critical for overall skeletal health and the prevention of osteoporosis. Post-menopausal women are at high risk of having osteoporosis and this risk is reduced when adequate VIT D status is maintained. VIT D is fat-soluble and only a limited number of foods naturally contain it. Also, while VIT D absorption is enhanced by dietary lipid, the optimal amount of lipid required for maximal absorption has not been determined. A paucity of data exists regarding the effect of a co-consumed food source of lipid to enhance VIT D absorption and the impact of aging on VIT D bioavailability in women.

ELIGIBILITY:
Inclusion Criteria:

* Pre- (regularly menstruating, aged 19-45y) and post-menopausal (aged 60+y) females
* weight stable (± 3 kg in the past 3 months)
* constant habitual activity patterns within last 3 months
* no acute illness
* not diabetic or have chronic diseases known to influence lipid or energy metabolism
* blood 25(OH)D>20 nmol/L
* non-smoking
* drinking no more than 2 alcoholic drinks per day
* not taking estrogen-based birth control or osteoporosis prevention or treatment medications in the past 3 months
* not taking lipid-lowering medications

Exclusion Criteria:

* Males
* age <19 or age >45y for pre-menopausal women and age <60y for post-menopausal women
* weight change>3 kg in the past 3 months
* exercising vigorously over the past 3 months
* intestinal disorders including lipid malabsorption or lactose intolerance
* abnormal liver or kidney function tests
* blood 25(OH)D<20 nmol/L
* fasting blood glucose>110 mg/dL
* smoking
* drinking more than 2 alcoholic drinks per day
* taking estrogen-based birth control or osteoporosis prevention or treatment medications in the past 3 months
* taking lipid-lowering medications affecting plasma cholesterol concentration

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Contents of total and individual carotenoids in triglyceride-rich lipoprotein fractions | From hour 0 to hour 10
  composite 0-10 h area under the curve of total and individual carotenoids (lutein, zeaxanthin, alpha-carotene, beta-carotene, lycopene) in triglyceride-rich lipoprotein fractions (all units are nmol/L x 10 hours)
Vitamin D content in in triglyceride-rich lipoprotein fractions | From hour 0 to hour 10
  composite 0-10 h area under the curve of vitamin D2, vitamin D3, 25(OH)D2, and 25(OH)D3 in triglyceride-rich lipoprotein fractions (all units are nmol/L x 10 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue Clinical Research Center, West Lafayette, Indiana, United States